CLINICAL TRIAL: NCT01309035
Title: Total Knee Arthroplasty - Accelerated Recovery Without Tourniquet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-001-AE
Record Dates: First submitted 2011-01-14; First posted 2011-03-04 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Arthropathy of Knee Joint
Keywords: Prothesis fixation; Bloodlessness
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With Tourniquet (Active Comparator): Total Knee Arthroplasty. Surgery performed during use of a tourniquet.
  Interventions: Procedure: Total Knee Arthroplasty
- Without Tourniquet (Experimental): Total Knee Arthroplasty. Surgery performed without use of a tourniquet.
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Surgery for OA knee pains

SUMMARY:
Introduction:

Approximately 7000 total knee replacements (TKAs) are done every year. More than 90% of these knee replacements are performed with the use of bone cement. Traditionally, a tourniquet has been, used to reduce the bleeding during surgery, enabling surgeons to perform delicate dissections in a bloodless operative field.

A tourniquet can be defined as a constricting or compressing device used to control temporarily venous and arterial circulation to an extremity. Pressure is applied circumferentially on the skin and underlying tissues of a limb. This pressure is transferred to the walls of vessels, causing them to become occluded.

It is well known that applying a tourniquet for more than 1 to 2 hours is associated with a number of disadvantages, for instance, severe pain and muscle effects during the first postoperative day, thereby slowing rehabilitation.

Other side effects related to tourniquet use, include pulmonary embolus caused by venous thrombosis and arterial thrombosis as a result of the dislodgement of an arterial plaque. Furthermore, tourniquet-induced hypertension with general anaesthesia, muscle injury, a wide spectrum of neurologic injuries, and tissue changes (Oedema compartment syndrome, post-tourniquet syndrome) have been reported. An important fact is that bleeding affects the quality of binding between bone and cement and thereby fixation of the knee prosthesis? Since the introduction of modern cementing techniques, no previous clinical studies have investigated the advantages or disadvantages of tourniquet use in knee replacement surgery.

Aims/hypothesis of the study:

1. To investigate the advantages and disadvantages of tourniquet use, including whether not using a tourniquet reduces pain, facilitates mobilisation and recovery, and shortens length of stay.
2. To study whether use of a tourniquet affects leg muscles during and after surgery, as measured by with use of microdialysis to quantify level of ischemia .
3. To determine whether prosthesis fixation, measured by RSA, is affected by tourniquet use. Because third generation cements secure prosthesis fixation, the investigators do not expect to find any clinically significant migration (less than 2 mm) 2 years after surgery.

Perspectives:

The investigators hope that the results of our study will improve rehabilitation regimes so that patients will experience less pain after surgery and thus achieve more rapid mobilisation and return to their daily lives.

DETAILED DESCRIPTION:
Design

Patients being able to participate in this study all have to fulfill the given inclusion criteria:

* Patients with symptomatic and radiographic verified knee symptoms, selected for primary unilateral total knee joint replacement (TKA)
* Age 50 and above (not older than 85)
* BMI < 35 and height >160 cm
* No severe cardiovascular conditions
* No previously knee surgery done in the same knee
* Oral and written acceptance

A group concerning 2 x 30 patients will be randomized into two groups. Either an intervention group, with absence of tourniquet or a control group with tourniquet. Which group they will belong to, is blinded to patient and surgeon until they reach operation room. The operation will be performed as usual, but with exception of two additional procedures. During operation small spheric tantalum pellets are placed around the prosthesis. Furthermore patients are prepared for microdialysis, which contain placement of 3 catheters: one in each thigh and one subcutaneously in the abdomen.

Microdialysis is a unique technique to monitor the chemistry of the extracellular space in living tissue. It is primarily used for In Vivo determinations of endogenous metabolites, thus serving as an indicator for ischemia.

RSA is precision radiology where the small pellets are visual on x-ray. Using computer a 3D image is created and the pellets serve as markers. These markers will be measured every 6 months showing whether a possible migration of the prosthesis is occurring and thereby indicating a loosening.

Out-patient treatment Patients will among other things be followed by clinical functional scores, registration of analgetica use, conventional X-ray and RSA In the long run the perspective is that surgery concerning knee replacements will be conducted without the use of tourniquet and thereby reducing the pain of the patients without compromising the end result of the operation, namely the fixation of the prosthesis.

Permissions approved by the Regional Committee on Biomedical Research Ethics, Region of Northern Jutland and Danish Data Protection Agency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic and radiographic verified knee symptoms, selected for primary unilateral total knee joint replacement (TKR)
* Age 50 and above (not older than 85)
* BMI < 35 and height >160 cm
* No severe cardiovascular conditions
* No previously knee surgery done in the same knee
* Oral and written acceptance

Exclusion Criteria:

* Severe obesity
* rheumatic diseases
* Absence of pulse in foot
* Diabetes
* Previous operation in concerning knee
* Lack of informed consent or ability to read / understand Danish

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Determine whether prosthesis fixation, measured by RSA, is affected by tourniquet use. | 1.Feb 2011 -1 jan 2013
  To determine whether prosthesis fixation, measured by RSA, is affected by tourniquet use. Because third generation cements secure prosthesis fixation, we do not expect to find any clinically significant migration (less than 2 mm) 2 years after surgery.

SECONDARY OUTCOMES:
To investigate the advantages and disadvantages of tourniquet use, including whether not using a tourniquet reduces pain, facilitates mobilisation and recovery, and shortens length of stay. | 1.feb 2011 - 1.jan 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Northern Orthopaedic Division, Department of Arthroplasty, Farsoe Clinic, Farsø, Northern Jutland, Denmark